CLINICAL TRIAL: NCT05386914
Title: Short Term Apolipoprotein E (ApoE)-Dependent Cerebral Blood Flow and Lung Perfusion Response to Sirolimus in Cognitively Normal Adults
Brief Title: Short Term Sirolimus Treatment and MRI of the Brain and Lungs
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Ai-Ling Lin, PhD, Professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2091042
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Genetic Predisposition to Disease; Healthy Volunteers
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carrier APOE4 (Experimental)
  Interventions: Drug: Sirolimus
- Non-Carrier APOE4 (Other)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 1 mg of Sirolimus taken orally once a day for 4 weeks.

SUMMARY:
Alzheimer's disease is a devastating neurodegenerative disease characterized by accumulation of clumps (also called plaques) and bundles of fibers (also called tangles) in the brain, for which there is currently no cure. Sirolimus is an FDA-approved medication which may improve the blood flow to the brain.

Part I: This study is designed to see if sirolimus treatment improves MRI blood flow to the brain in individuals with and without a genetic predisposition to Alzheimer's disease. Part I of this study is complete and no longer enrolling participants.

Part II: Ongoing research will expand the genetic predisposition cohort and further explore the drug's impact on the lung perfusion via hyperpolarized xenon-129 gas MRI and the brain-vascular connection. Only subjects who are APOE4 carriers will be enrolled in Part II.

Hyperpolarized xenon-129 gas MRI is a non-invasive technique in which a subject inhales a bolus of hyperpolarized xenon-129 gas which can be directly imaged by the MRI as it physiologically distributes itself throughout the lung interior and within tissue and red blood cells. It thus allows for direct imaging and quantification of regional lung function: ventilation, gas-exchange, and perfusion. The relationship between pulmonary vascular function and brain perfusion is largely unstudied. We hope to investigate the relationship between pulmonary vascular function and cerebral blood flow by quantifying both lung and brain perfusion before and after the administration of Sirolimus.

ELIGIBILITY:
Part I:

Inclusion Criteria:

* 1. Age 45-65 y/o
* 2. Male or female, all ethnic groups
* 3. Montreal Cognitive Assessment (MoCA) score greater than or equal to 26
* 4. Clinical Dementia Rating (CDR) Staging Instrument = 0
* 5. Carrier Cohort: APOE4 homozygous or heterozygous
* 6. Non-Carrier cohort: no APOE4 gene identified

Exclusion Criteria:

* 1. Diagnosis of mild cognitive impairment (MCI) or dementia, including Alzheimer's disease
* 2. BMI ≥35 (based on MRI feasibility)
* 3. Diabetes (HBA1c≥6.5% or antidiabetic medications)
* 4. History of skin ulcers or poor wound healing
* 5. Current tobacco or illicit drug use or alcohol abuse (defined as ≥4 per day or ≥14 per week for men and ≥3 per day or ≥7 per week for women) (Per NIAAA guidelines)
* 6. Use of anti-platelet or anti-coagulant medications other than aspirin
* 7. Current medications that affect cytochrome P450 3A4 (CYP3A4)
* 8. Immunosuppressant therapy within the last year
* 9. Chemotherapy or radiation treatment within the last year
* 10. Current or chronic history of liver or kidney disease or known hepatic or biliary abnormalities
* 11. Untreated hypertriglyceridemia (fasting triglycerides < 300 mg/dl)
* 12. Current or chronic significant history of pulmonary disease
* 13. Chronic heart failure
* 14. Pregnancy or lactation
* 15. Recent history (past six months) of myocardial infarction, active coronary artery disease, intestinal disorders, stroke, or transient ischemic attack
* 16. Poorly controlled blood pressure (systolic BP>160 or diastolic BP>100 mmHg)
* 17.Active inflammatory, Coronavirus (COVID-19), autoimmune, infectious, hepatic, gastrointestinal, malignant, and/or severe mental illness
* 18. History of, or MRI, or CT positive for, any space occupying brain lesion, including mass effect or abnormal intracranial pressure
* 19. Organ transplant recipients
* 20. History of Stroke
* 21. History of ruptured intracranial aneurysm
* 22. Any condition for which a MRI procedure is contraindicated. Some examples include: metallic material in the body, such as pacemakers, metallic clips, etc.
* 23. Likelihood of claustrophobia

Part II:

The inclusion and exclusion criteria for Part I apply to Part II with the addition of the following:

Exclusion Criteria:

1. Baseline oxygen requirement
2. Blood oxygen saturation of 90% or less than as measured by pulse oximetry on the day of imaging
3. FEV1 percent predicted less than 25%
4. Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in the eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded
5. Chest circumference greater than that of the xenon-129 MR coil. The circumference of the coil is approximately 42 inches
6. History of congenital cardiac disease or history of apneic episodes
7. Inability to understand simple instructions or to hold still for approximately 10 seconds
8. History of respiratory infection within 2 weeks prior to the MR scan

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow as measured on MRI | Baseline to 4 weeks
  Rate of blood perfusion expressed as mL/100g/min globally and regionally

SECONDARY OUTCOMES:
Part I: Plasma and Microbiome Biomarkers | Part I: Baseline to 4 weeks
  Part I: To assess baseline-to-post-treatment changes in plasma metabolomics and short-chain-fatty-acids (SCFA) profiles
Part I: Plasma and Microbiome Markers | Part I: Baseline to 4 weeks
  Part I: To assess baseline-to-post-treatment changes in plasma markers associated with AD pathology
Part I: Plasma and Microbiome Biomarkers | Part I: Baseline to 4 weeks
  Part I: To assess baseline-to-post-treatment changes in plasma cytokine levels
Part I: Plasma and Microbiome Markers | Part I: Baseline to 4 weeks
  Part I: To assess baseline-to-post-treatment gut microbiome diversity and composition
Part II: RBC/Membrane Ratio | Part II: Baseline to 4 weeks
  Part II: In addition to the outcome measures listed for Part I of this study, the secondary outcome measures for Part II are as follows: ratio of xenon signal dissolved in RBCs to xenon signal dissolved in membrane tissues

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Ling Lin, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ficke AJ, Owens WF Jr. Femoral shaft fractures and the above-knee amputee: use of the compression plate. A report of three cases. Clin Orthop Relat Res. 1972 Sep;87:200-3. No abstract available. PMID 4562190
- [Background] Abstracts. Metastasis Congress. Heidelberg, September 26-29, 1988. 2nd international conference. Clin Exp Metastasis. 1988;6 Suppl 1:1-99. No abstract available. PMID 3409562
- [Background] Lynch T, Price A. The effect of cytochrome P450 metabolism on drug response, interactions, and adverse effects. Am Fam Physician. 2007 Aug 1;76(3):391-6. PMID 17708140
- [Background] Kraig E, Linehan LA, Liang H, Romo TQ, Liu Q, Wu Y, Benavides AD, Curiel TJ, Javors MA, Musi N, Chiodo L, Koek W, Gelfond JAL, Kellogg DL Jr. A randomized control trial to establish the feasibility and safety of rapamycin treatment in an older human cohort: Immunological, physical performance, and cognitive effects. Exp Gerontol. 2018 May;105:53-69. doi: 10.1016/j.exger.2017.12.026. Epub 2018 Feb 3. PMID 29408453
- [Background] Ozcelik S, Fraser G, Castets P, Schaeffer V, Skachokova Z, Breu K, Clavaguera F, Sinnreich M, Kappos L, Goedert M, Tolnay M, Winkler DT. Rapamycin attenuates the progression of tau pathology in P301S tau transgenic mice. PLoS One. 2013 May 7;8(5):e62459. doi: 10.1371/journal.pone.0062459. Print 2013. PMID 23667480
- [Background] Spilman P, Podlutskaya N, Hart MJ, Debnath J, Gorostiza O, Bredesen D, Richardson A, Strong R, Galvan V. Inhibition of mTOR by rapamycin abolishes cognitive deficits and reduces amyloid-beta levels in a mouse model of Alzheimer's disease. PLoS One. 2010 Apr 1;5(4):e9979. doi: 10.1371/journal.pone.0009979. PMID 20376313
- [Background] Ross C, Salmon A, Strong R, Fernandez E, Javors M, Richardson A, Tardif S. Metabolic consequences of long-term rapamycin exposure on common marmoset monkeys (Callithrix jacchus). Aging (Albany NY). 2015 Nov;7(11):964-73. doi: 10.18632/aging.100843. PMID 26568298
- [Background] Tardif S, Ross C, Bergman P, Fernandez E, Javors M, Salmon A, Spross J, Strong R, Richardson A. Testing efficacy of administration of the antiaging drug rapamycin in a nonhuman primate, the common marmoset. J Gerontol A Biol Sci Med Sci. 2015 May;70(5):577-87. doi: 10.1093/gerona/glu101. Epub 2014 Jul 19. PMID 25038772
- [Background] Sills AM, Artavia JM, DeRosa BD, Ross CN, Salmon AB. Long-term treatment with the mTOR inhibitor rapamycin has minor effect on clinical laboratory markers in middle-aged marmosets. Am J Primatol. 2019 Feb;81(2):e22927. doi: 10.1002/ajp.22927. Epub 2018 Oct 12. PMID 30311681
- [Background] Lelegren M, Liu Y, Ross C, Tardif S, Salmon AB. Pharmaceutical inhibition of mTOR in the common marmoset: effect of rapamycin on regulators of proteostasis in a non-human primate. Pathobiol Aging Age Relat Dis. 2016 Jun 23;6:31793. doi: 10.3402/pba.v6.31793. eCollection 2016. PMID 27341957
- [Background] Lin AL, Parikh I, Yanckello LM, White RS, Hartz AMS, Taylor CE, McCulloch SD, Thalman SW, Xia M, McCarty K, Ubele M, Head E, Hyder F, Sanganahalli BG. APOE genotype-dependent pharmacogenetic responses to rapamycin for preventing Alzheimer's disease. Neurobiol Dis. 2020 Jun;139:104834. doi: 10.1016/j.nbd.2020.104834. Epub 2020 Mar 12. PMID 32173556
- [Background] Lin AL, Jahrling JB, Zhang W, DeRosa N, Bakshi V, Romero P, Galvan V, Richardson A. Rapamycin rescues vascular, metabolic and learning deficits in apolipoprotein E4 transgenic mice with pre-symptomatic Alzheimer's disease. J Cereb Blood Flow Metab. 2017 Jan;37(1):217-226. doi: 10.1177/0271678X15621575. Epub 2015 Dec 31. PMID 26721390
- [Background] Lin AL, Zheng W, Halloran JJ, Burbank RR, Hussong SA, Hart MJ, Javors M, Shih YY, Muir E, Solano Fonseca R, Strong R, Richardson AG, Lechleiter JD, Fox PT, Galvan V. Chronic rapamycin restores brain vascular integrity and function through NO synthase activation and improves memory in symptomatic mice modeling Alzheimer's disease. J Cereb Blood Flow Metab. 2013 Sep;33(9):1412-21. doi: 10.1038/jcbfm.2013.82. Epub 2013 Jun 26. PMID 23801246
- [Background] Mannick JB, Del Giudice G, Lattanzi M, Valiante NM, Praestgaard J, Huang B, Lonetto MA, Maecker HT, Kovarik J, Carson S, Glass DJ, Klickstein LB. mTOR inhibition improves immune function in the elderly. Sci Transl Med. 2014 Dec 24;6(268):268ra179. doi: 10.1126/scitranslmed.3009892. PMID 25540326